CLINICAL TRIAL: NCT07269639
Title: Golcadomide, Poseltinib, and Rituximab for Optimized Treatment of Relapsed/Refractory Diffuse Large B-cell Lymphoma (Go-Pro-DLBCL)
Brief Title: Golcadomide, Poseltinib, and Rituximab for Relapsed/Refractory Diffuse Large B-cell Lymphoma
Acronym: Go-Pro-DLBCL
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, JaMin Byun, M.D. Ph.D., Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-2507-184-1662
Record Dates: First submitted 2025-11-25; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Large B-Cell Lymphoma (LBCL)
Keywords: large b-cell lymphoma; golcadomide; poseltinib; rituximab
MeSH Terms: interventions — poseltinib; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment arm (Experimental): golcadomide + poseltinib + rituximab (GoPro)
  Interventions: Drug: Golcadomide + Poseltinib + Rituximab

INTERVENTIONS:
Drug: Golcadomide + Poseltinib + Rituximab — Participants will receive 0.4 mg of golcadomide once daily for 14 consecutive days for 18 cycles in 28-day cycles. The first 6 cycles will be administered in combination with rituximab and poseltinib, while the remaining 12 cycles will be conducted with poseltinib alone. During the maintenance period (Cycles 7-18), the first day of study treatment administration with golcadomide is designated as Day 1 of each cycle.
  Rituximab can be administered with or up to 2 hours after the morning dose of golcadomide in the fed or fasted state. For Cycles 1-6, the first day of study treatment administration with rituximab is designated as Day 1 of each cycle. Rituximab will be administered as an IV infusion at a dose of 375 mg/m2 on Days 1, 8, 15, and 22 of Cycle 1, and Day 1 of Cycles 2-6.
  Poseltinib is administered orally twice daily, approximately every 12 hour. Part 1 (safety cohort) of the study will be conducted in up to approximately 9 participants to select the optimal RP2D of poseltinib.

SUMMARY:
This trial is a proof-of-concept, pilot study, phase I/II clinical trial aimed at generating preliminary data on the combination of golcadomide, poseltinib, and rituximab.

DETAILED DESCRIPTION:
This is a single arm, open-label, phase I/II trial of Poseltinib in combination with golcadomide and rituximab in patients with relapsed or refractory diffuse large B-cell lymphoma. Considering (1) the combination of BTK inhibitor, lenalidomide, and rituximab has demonstrated efficacy in R/R DLBCL, (2) golcadomide, a CELMoD, exhibits potent immunomodulatory activity compared to IMiDs such as lenalidomide, and (3) poseltinib is a potent, covalent BTK inhibitor with more than twice the selectivity for BTK compared to other BTK inhibitors, we anticipate that this combination will yield promising results in R/R DLBCL.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must satisfy the following criteria to be enrolled in the study

  1. Subject is ≥ 19 years of age at the time of signing the informed consent form (CRF).
  2. Subject must understand and voluntarily sign an ICF prior to any study-related assessments/procedures being conducted.
  3. Subject is willing and able to adhere to the study visit schedule and other protocol requirements.
  4. Subject has histologically confirmed (per local evaluation) diagnosis of aggressive large B-cell lymphoma according to 2022 WHO classification, specifically:

     A. DLBCL, NOS (including GCB and ABC types) B. DLBCL/high grade B-cell lymphoma, with MYC and BCL2 rearrangements C. High grade B-cell lymphoma, NOS D. T-cell/histiocyte-rich large B-cell lymphoma E. EBV-positive DLBCL
  5. Relapsed or refractory disease following at least 1 prior line of therapy (must include an anthracycline-based treatment), and ineligible for hematopoietic stem cell transplantation.
  6. Subjects must have measurable disease defined by at least one fluorodeoxyglucose (FDG)-avid lesion for FDG-avid subtype and one bi-dimensionally measurable (> 1.5 cm in longer diameter) disease by computed tomography (CT) or magnetic resonance imaging (MRI), as defined by the Lugano classification.
  7. Subject has an Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.
  8. Subject must have the following laboratory values:

     A. ANC ≥ 1.0 × 109/L or ≥ 0.5 × 109/L in case of documented bone marrow involvement of DLBCL-related hypersplenism present. It is not permissible to administer G-CSF to achieve minimum ANC levels within 7 days prior to screening complete blood count (or within 14 days prior for pegfilgrastim).

     B. Hemoglobin ≥ 75 g/L (7.5 g/dL). Transfusion is permitted in cases of bone marrow involvement of lymphoma, and screening will be conducted at least one week after transfusion.

     C. Platelets ≥ 75 × 109/L or ≥ 50 × 109/L in case of documented bone marrow involvement of DLBCL-related hypersplenism present, without transfusion for 7 days.

     D. AST and ALT ≤ 2.5 × ULN. In case of documented liver involvement by lymphoma, AST and ALT must be ≤ 5.0 × ULN.

     E. Serum total bilirubin ≤ 1.5 × ULN (corresponding to mild dysfunction as per National Cancer Institute Organ Dysfunction Working Group [NCI ODWG] criteria). In case of documented liver involvement by lymphoma, serum total bilirubin must be ≤ 3.0 × ULN.

     F. Estimated serum CrCL of ≥ 30 mL/min using the modification of diet in renal disease (MDRD) formula G. International normalized ratio (INR) < 1.5 × ULN and activated partial thromboplastin time (aPTT) < 1.5 × ULN (for subjects not receiving therapy). Note: subjects receiving therapy for a thromboembolic event that occurred > 3 months prior to enrollment are eligible as long as they are on a stable regimen of anticoagulation with warfarin, low-molecular weight heparin, or other approved therapeutic anticoagulation or antiplatelet regimen.
  9. Individual of childbearing potential (IOCBP) must:

     A. Have two negative pregnancy tests as verified by the investigator prior to starting study treatment. She must agree to ongoing pregnancy testing during the course of the study, and after the end of study treatment. This applies even if the subject practices true abstinence* from heterosexual contact.

     B. Either commit to true abstinence* from heterosexual contact (which must be reviewed on a monthly basis and source documented) or agree to use, and be able to comply with, 2 forms of contraception: one highly effective, and one additional effective (barrier) measure of contraception without interruption 28 days prior to starting study treatment, during the study treatment (including dose interruptions), and for at least 28 days after the last dose of golcadomide, and for 12 months after the last dose of rituximab and poseltinib, whichever is longer.

     Note: IOCBP is an individual who: 1) has achieved menarche (first menstrual cycle) at some point; 2) has not undergone a hysterectomy (the surgical removal of the uterus) or bilateral salpingectomy (the surgical removal of the fallopian tubes) or oophorectomy (the surgical removal of both ovaries) or 3) has not been naturally postmenopausal (without an alternative medical cause, e.g. amenorrhea following cancer therapy does not rule out childbearing potential) for at least 12 consecutive months (ie, has had menses at any time during the preceding 12 consecutive months).
  10. Female subjects must agree to refrain from donating eggs while on study treatment and for at least 28 days after last dose of golcadomide.
  11. Male subjects must:

      A. Practice true abstinence* (which must be reviewed on a monthly basis) or agree to use a condom during sexual contact with a pregnant individual or an IOCBP while participating in the study, during dose interruptions, and for at least 28 days after the last dose of golcadomide or 90 days for rituximab or 12 months for poseltinib, whichever is longer, even if he has undergone a successful vasectomy.

      B. Agree to refrain from donating sperm or semen while on study treatment, during dose interruptions and for at least 12 months after last dose of study treatment.

      * True abstinence is acceptable when this is in line with the preferred and usual lifestyle of the subject. [Periodic abstinence (e.g., calendar, ovulation, post-ovulation methods) and withdrawal are not acceptable methods of contraception].
  12. Subjects must:

A. Agree to refrain from donating blood while on study treatment, during dose interruptions and for at least 28 days following the last dose of golcadomide.

B. Agree to refrain from receiving live vaccines while on study treatment, during dose interruptions and for at least 90 days following the last dose of the study treatment.

C. Agree not to share study medication with another person.

Exclusion Criteria:

* The presence of any of the following will exclude a subject from enrollment:

  1. Subject who has had prior treatment with golcadomide.
  2. Subject who has had prior treatment with BTK inhibitor.
  3. Subject has life expectancy ≤ 2 months.
  4. Subject has received any of the following:

     A. Major surgery (as defined by the Investigator) within 28 days of initiating study treatment. Subjects must have recovered from any clinically significant effects of recent surgery.

     B. Radiation therapy within 28 days prior to initiating study treatment. C. Use of any systemic anti-cancer treatment (approved or investigational) within 28 days or 5 half-lives prior to starting study treatment, whichever is shorter. (Participation in another interventional clinical trial concurrent with this study is not permitted, except for those who have completed treatment with the prior investigational agent(s) and are currently in long-term follow up)
  5. Subject has previously received solid organ transplantation.
  6. Subject has undergone allogeneic SCT within 1 year prior to initiating study treatment or autologous SCT within 3 months prior to initiating study treatment.

     A. Subject who had received prior SCT should not have any Grade >1 treatment-related toxicity.

     B. Subject who had received prior SCT should not have clinically significant, active graft-versus-host disease (GVHD).
  7. Subject has any other subtype of lymphoma. Cases of primary mediastinal (thymic) large B-cell lymphoma, primary cutaneous DLBCL-leg type, Grade 3b FL, ALK-positive large B-cell lymphoma, primary effusion lymphoma, or Burkitt lymphoma are excluded.
  8. Subject has active central nervous system (CNS) involvement by lymphoma
  9. Subject has any significant medical condition (e.g., uncontrolled diabetes mellitus, uncontrolled hypertension), including active or uncontrolled infection, presence of laboratory abnormality, or psychiatric illness that places the subject at an unacceptable risk for treatment-related complications, if he/she were to participate in the study.
  10. Subject has any condition that confounds the ability to interpret data from the study.
  11. Persistent diarrhea or malabsorption grade ≥ 2 NCI CTCAE, despite medical management. Subject with gastrointestinal disease or surgery (e.g., gastric bypass surgery) that may significantly alter the absorption of oral study treatment.
  12. Subject has a prior history of malignancies other than lymphoma, except if the participant has been free of the disease for at least 3 years. Exceptions to the ≥ 3-year time limit include history of the following:

      A. Localized nonmelanoma skin cancer B. Carcinoma in situ of the cervix C. Carcinoma in situ of the breast D. Incidental histologic finding of prostate cancer (T1a or T1b as per Tumor Node Metastasis staging system) or prostate cancer that has been treated with curative intent
  13. Subject has impaired cardiac function or clinically significant cardiovascular disease, defined as any of the following within 6 months prior to enrollment:

      A. Acute myocardial infarction or acute coronary syndromes (e.g., unstable angina, coronary artery bypass graft, coronary angioplasty or stenting, symptomatic pericardial effusion) B. Clinically significant cardiac arrhythmias (e.g., uncontrolled atrial fibrillation, uncontrolled paroxysmal supraventricular tachycardia, persistent ventricular arrhythmias) C. Prolonged QT syndrome (or QTcF ≥ 470 msec on screening electrocardiogram) D. Left ventricular ejection fraction (LVEF) < 45% as determined by multigated acquisition scan (MUGA) or echocardiogram (ECHO) E. Complete left bundle branch or bifascicular block
  14. Concurrent administration of strong CYP3A4/5 modulators. The washout period for strong CYP3A4/5 modulators is 7 days or 5 half-lives (whichever is longer) before initiation of golcadomide.
  15. Subject is unable or unwilling to undergo protocol required thromboembolism or antiviral prophylaxis.
  16. Subject is positive for human immunodeficiency virus (HIV), chronic or active hepatitis B, active hepatitis A, or active hepatitis C:

      A. Known positive HIV status B. Seropositive for hepatitis B (defined by a positive test for hepatitis B surface antigen [HBsAg] either acute or chronic hepatitis). Subjects with resolved infection (i.e., subjects who are HBsAg negative but positive for antibodies to hepatitis B core antigen [anti-HBcAb] and/or antibodies to hepatitis B surface antigen [anti-HBsAb]) must be screened using real-time polymerase chain reaction (PCR) measurement of HBV deoxyribonucleic acid (DNA) levels. Those who are PCR positive will be excluded. HBV carriers without active disease (HBV DNA titer < 1000 copies/mL or 200 IU/mL) may be enrolled in the study with adequate anti-viral prophylaxis.

      EXCEPTION: Subjects with serologic findings suggestive of HBV vaccination (anti-HBs positivity as the only serologic marker) AND a known history of prior HBV vaccination, do not need to be tested for HBV DNA by PCR.

      EXCEPTION: Subjects with positive anti-HBcAb but negative HBsAg and negative anti-HBsAb profiles are eligible if HBV DNA PCR is negative.

      C. Known to be seropositive for hepatitis C virus (HCV); anti-HCV antibody positive and HCV- ribonucleic acid (RNA) quantitation positive. Cured HCV patients (negative for HCV RNA test) may be enrolled in the study.
  17. Subject hast a history of anaphylaxis or hypersensitivity to investigational products or components of investigational products (rituximab, golcadomide, poseltinib).
  18. Subject is an individual who is pregnant, nursing, or breastfeeding, or who intends to become pregnant during participation in the study.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | The evaluation time frame is from baseline up to 18 months.
  The primary endpoint was the Overall response rate, defined as the proportion of participants who achieved either CMR or PMR according to the Lugano criteria 2014. The primary analysis will be conducted in the efficacy evaluable population.
  A one-sample exact binomial test (one-sided, α=0.05) will be used to compare the observed ORR against the null hypothesis value of 30%. If the lower bound of the exact one-sided 95% CI for the observed ORR exceeds 30%, the null hypothesis will be rejected, suggesting that the combination therapy demonstrates meaningful efficacy.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | The evaluation time frame extends from baseline to 1 year and 3 year after the last patient in.
  PFS is calculated as the time from enrollment to the first documented progression confirmed or death due to any cause, whichever occurs first. Response assessments will be based on the Lugano criteria 2014. PFS analysis will follow the censoring rules based on Food and Drug Administration (FDA) guideline (2018) as the primary analysis method. Specifically, subjects who initiated other anti-lymphoma therapy without documented PD will be censored at last adequate assessment prior to the initiation of other anti-lymphoma therapy. Subjects with two or more consecutive missed assessments prior to documented PD or death will be censored at the last adequate assessment prior to the missing assessment. The Kaplan-Meier method will be used to estimate the survival distribution functions. The median PFS along with the two-sided 95% CI for the median will be estimated.
Overall survival (OS) | The evaluation time frame extends from baseline to 3 years after the last patient in.
  OS is calculated as the time from randomization to death from any cause. Subjects who died will be considered as having OS events on the date of death. All subjects who are lost to follow-up prior to the date of the data cut-off or who withdrew consent from the trial will be censored at the last date known to be alive. Subjects who are still in the study at the date of data cut-off will be censored at the last available date that the subject is known to be alive, or data cut-off date, whichever is earlier. The analysis of OS will be based on all data available. The median OS along with the two-sided 95% confidence interval for the median will be estimated.
Complete metabolic response (CMR) rate | The evaluation time frame is from baseline up to 18 months.
  The CMR rate is the proportion of subjects who achieve CMR according to the Lugano criteria 2014.
Duration of response (DOR) | The evaluation time frame extends from baseline to 1 year and 3 years after the last patient in.
  DoR is calculated as the time from first documentation of response (CMR or PMR) to the first documented progression confirmed, start of new anti-lymphoma therapy, or death due to any cause, whichever occurs first. Response assessments will be based on the Lugano criteria 2014. The analysis will be conducted in patients who achieved a documented response. The Kaplan-Meier method will be used to estimate the survival distribution functions for each treatment arm. The median DoR along with the two-sided 95% confidence interval for the median will be estimated.
Recommended poseltinib dose | through study part 1 completion, up to 8 weeks.
  In Part 1 (safety cohort; dose-finding phase), the recommended poseltinib dose for Part 2 will be determined based on the totality of safety and efficacy data, selecting between 40 mg BID and 60 mg BID.
Safety | from C1D1 to end of trial, assessed up to 3 years after the last patient in.
  Safety data will be summarized for the safety cohort. The baseline value for the safety analysis is defined as the value collected at the time closest to and before the start of study intervention administration. Estimates of safety measures (adverse events) will be summarized with frequency (%).

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided